CLINICAL TRIAL: NCT05963061
Title: Chronic Myeloid Leukemia (CML) Real-Life Database
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Centre Hospitalier Universitaire de Saint Etienne (Other); Bicetre Hospital (Other); University Hospital, Caen (Other); Central Hospital, Nancy, France (Other); University Hospital, Toulouse (Other); CH Annecy Genevois (Other); Rennes University Hospital (Other); Hopital Paul Brousse (Other); Versailles Hospital (Other); Centre Hospitalier Emile Roux (Other); University Hospital, Limoges (Other); Institut Paoli-Calmettes (Other); Centre Hospitalier de Rochefort (Other)
Responsible Party: Sponsor
Other Study IDs: CML Observatory
Record Dates: First submitted 2023-02-20; First posted 2023-07-27 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-02

CONDITIONS: Chronic Myeloid Leukemia (CML)
Keywords: Leukemia; Leukemia, Myeloid; Chronic myeloid leukemia; Chronic, BCR::ABL Positive; Hematologic Malignancies; Tyrosine kinase inhibitor (TKI); Targeted therapy
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Leukemia; Leukemia, Myeloid; Bronchiolitis Obliterans Syndrome; Hematologic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 30 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Establish the largest possible real-life cohort collecting long-term follow-up of a maximum number of CML patients in order to carry out observational studies: epidemiological, identification of subgroups according to their response to treatment, evaluation of new molecules in real life, therapeutic discontinuations, impact of the evolution of recommendations, etc.

DETAILED DESCRIPTION:
Observational study collecting real-life clinico-biological data from patients with CML. Data are collected prospectively and retrospectively, from diagnosis and throughout the long-term follow-up of CML (follow up continues after treatment stopped).

ELIGIBILITY:
Inclusion Criteria:

* Patient diagnosed for chronic myelocytic leukemia

Exclusion Criteria:

* CML allograft without TKI treatment
* Refusal or inability to sign the consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Any patient with a diagnose of CML
Sampling Method: Non-Probability Sample
Enrollment: 3500 (Estimated)
Dates: Start 2014-04-16 (Actual); Primary Completion 2034-04-16 (Estimated); Study Completion 2034-04-16 (Estimated)

PRIMARY OUTCOMES:
Clinical and biological data collection | Until death or last follow up (up to 30 years)
  Aims of the registry are the collection of clinical data to gain further insights about patients's CML treated with ITK's (treatment, prognosis, therapeutical response).

SECONDARY OUTCOMES:
Prognosis score for CML (Sokal, ELTS, Eutos, Hasford) | At diagnosis
BMI with evaluation of weight and height | Until death or last follow up (up to 30 years)
Evaluation of major molecular response (MMR) with transcript BCR::ABL in % | Until death or last follow up (up to 30 years)
Evaluation of molecular response MR4 with transcript BCR::ABL in % | Until death or last follow up (up to 30 years)
Evaluation of molecular response MR4.5 with transcript BCR::ABL in % | Until death or last follow up (up to 30 years)
Evaluation of molecular response MR5 with transcript BCR::ABL in % | Until death or last follow up (up to 30 years)
Evaluation of cytogenetic response | Until death or last follow up (up to 30 years)
Evaluation of TKI efficacy based on transcript BCR::ABL in % | Until death or last follow up (up to 30 years)
Evaluation of TKI tolerance (adverses events) | Until death or last follow up (up to 30 years)
Calcul in month of the duration of maintenance TFR (treatment free remission) after stop TKI for thérapeutic response | Until death or last follow up (up to 30 years)
Listing of major medical history of patient's CML | Until death or last follow up (up to 30 years)

CONTACTS AND LOCATIONS:
Overall Officials: Marc BERGER, MD, Study Director — University Hospital, Clermont-Ferrand
Locations (14):
- France (14):
  - CH Annecy Genevois, Annecy
  - University Hospital, Caen, Caen
  - CHU Clemront-Ferrand, Clermont-Ferrand
  - Centre Hospitalier Emile Roux, Le Puy-en-Velay
  - University Hospital, Limoges, Limoges
  - Institut Paoli-Calmettes, Marseille
  - Centre Hospital, Nancy, Nancy
  - Bicetre Hospital, Paris
  - Hopital Paul Brousse, Paris
  - Rennes University Hospital, Rennes
  - Centre Hospitalier de Rochefort, Rochefort
  - Centre Hospitalier Universitaire de Saint Etienne, Saint-Etienne
  - University Hospital, Toulouse, Toulouse
  - Versailles Hospital, Versailles

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Saugues S, Lambert C, Daguenet E, Ansah HJ, Turhan A, Huguet F, Guerci-Bresler A, Tchirkov A, Hamroun D, Hermet E, Pereira B, Berger MG. Real-world therapeutic response and tyrosine kinase inhibitor discontinuation in chronic phase-chronic myeloid leukemia: data from the French observatory. Ann Hematol. 2022 Oct;101(10):2241-2255. doi: 10.1007/s00277-022-04955-z. Epub 2022 Aug 30. PMID 36040480
- See also: Real-world therapeutic response and tyrosine kinase inhibitor discontinuation in chronic phase-chronic myeloid leukaemia: Data from the French observatory — https://link.springer.com/article/10.1007/s00277-022-04955-z